CLINICAL TRIAL: NCT00446173
Title: Autologous Purged Hematopoietic Stem Cell Transplantation for Chronic Myelogenous Leukemia (CML)
Brief Title: Autologous Stem Cell Transplants for Chronic Myelogenous Leukemia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to low accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Marcos de Lima, MD/Associate Professor, U.T.M.D. Anderson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003-0710
Record Dates: First submitted 2007-03-09; First posted 2007-03-12 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Leukemia
Keywords: Chronic Myelogenous Leukemia; Leukemia; Philadelphia (Ph) chromosome positive CML; Busulfan; Busulfex; Myleran; Cyclophosphamide; Cytoxan; Neosar; G-CSF; Filgrastim; Neupogen; GM-CSF; Sargramostim; Leukine
MeSH Terms: conditions — Leukemia; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Busulfan; Cyclophosphamide; Granulocyte Colony-Stimulating Factor; Filgrastim; Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Busulfan + Cyclophosphamide + G-CSF + GM-CSF (Experimental)
  Interventions: Drug: Busulfan; Drug: Cyclophosphamide; Drug: G-CSF; Drug: GM-CSF

INTERVENTIONS:
Drug: Busulfan — 130 mg/m^2 IV Daily Over 3 Hours x 4 Days
  Other Names: Bulsulfex; Myleran
Drug: Cyclophosphamide — 60 mg/kg IV Daily Over 4 Hours x 2 Days
  Other Names: Cytoxan; Neosar
Drug: G-CSF — 10 mcg/kg Subcutaneously Once Daily
  Other Names: Filgrastin; Neupogen
Drug: GM-CSF — 250 mcg/kg Subcutaneously Once Daily
  Other Names: Sargramostim; Leukine

SUMMARY:
Primary Objective:

1. To study ex-vivo purging of autologous hematopoietic stem cells that will be used to support high-dose chemotherapy in patients with chronic myelogenous leukemia (CML). Major endpoints are neutrophil engraftment and survival.

Secondary Objectives:

1. To evaluate the toxicity of ex-vivo purged autologous cells when used to support high-dose chemotherapy.
2. To evaluate the rate and duration of cytogenetic remissions achieved with this strategy.
3. To determine the time to platelet recovery to 20,000/mm3.
4. To determine the one-year survival rate.

DETAILED DESCRIPTION:
Before treatment starts, you will have a complete physical exam. You will have about 4 tablespoons of blood drawn for tests to check on the status of the disease, to check organ functions, and to check for infectious diseases (hepatitis, HIV, etc.). You will have a sample of bone marrow collected. To collect a bone marrow sample, an area of the hip or chest bone is numbed with anaesthetic and a small amount of bone marrow is withdrawn through a large needle. You will also have heart (cardiac ejection fraction) and lung function tests. All of these tests are being done to make sure you are eligible for this treatment.

In order to access the blood in the circulation, a silicone catheter (small plastic tube) will be placed in the collar bone area. You will be under local anesthesia during this procedure. If you are found to be eligible to take part in this study, this catheter will be used for the collection of stem cells, infusion of chemotherapy, fluids, electrolytes, other medications, and also for blood sampling for lab tests. It will remain in your body for the length of the treatment (between 2-5 months).

Normally, there are very few stem cells in the blood. The majority of them are in the bone marrow. To help move or "mobilize" the cells needed from your bone marrow to your blood, you will be given chemotherapy followed by injections under the skin once a day of a drug called G-CSF and another drug called GM-CSF. These injections will be given over 7-21 days. The injections may be given by a nurse in the hospital, in the outpatient setting, or you may learn how to give them to yourself.

The chemotherapy you will receive to help mobilize the stem cells is cyclophosphamide. It will be given by vein over a few hours in one day. This is the first step toward collecting the stem cells necessary for transplantation later on. It is separate from the high-dose chemotherapy that you get after the transplant.

Blood samples (about 4 teaspoons each) will be drawn once a day after the cyclophosphamide to check for the numbers of stem cells in your blood and to monitor for possible side effects. If the number of stem cells in the blood is high enough, you will go to the UTMDACC Apheresis Unit and have your peripheral blood progenitor cells (PBPC, or stem cells) collected.

The procedure to collect your cells is called leukapheresis. It is similar to donating platelets to a blood bank. The cells will be removed from the blood through the catheter and the remaining blood will be given back to you through the catheter. This procedure is performed in a machine that processes the blood and separates the cells needed for transplantation, giving the rest back to you. Each leukapheresis procedure takes about 4-6 hours. You will have one leukapheresis procedure a day, for 1 to 5 days in a row, until enough stem cells are collected for the transplant and for ""back-up" in case of problems with the treated cells. If after 5 procedures, the number of cells collected is too low, additional collections of cells may be needed.

Some people may not be able to have enough cells collected through the blood. If this is the case, you may need to have bone marrow stem cells collected. You will be taken to the operating room and have multiple collections of bone marrow performed. The procedure will be performed while you are under general anesthesia. About 1 - 1.5 liters of bone marrow will be collected. You will be asked to donate your own blood before the procedure if possible. That blood will be given back to you in the operating room. Somebody else's blood may be given to you instead if you cannot donate.

After enough stem cells are collected, the cells will be treated in the laboratory, using Gleevec (imatinib mesylate) followed by ex vivo culture/purging. Culture-purging is a method that takes advantage of the fact that CML cells die when kept in laboratory culture in a shorter time period than normal blood cells. If the cells are kept alive long enough, surviving cells will be less contaminated by CML cells. Imatinib mesylate will provide a chemical way of killing the CML cells, since they are more toxic to CML cells than they are to normal cells. The culture-purging will also use three medications called "growth factors". The medications being used are stem cell factor, G-CSF, and thrombopoietin.

Busulfan and cyclophosphamide are chemotherapy drugs that are designed to kill leukemia cells. However, the combination will kill a significant amount of your bone marrow cells, which will basically stop the production of blood components. In order to restart the production, the cells that were removed and treated in the lab will be given back to you (autologous transplant).

You will be admitted to the hospital to receive high dose chemotherapy. You will be given busulfan by continuous injection (using the catheter) for 4 days, then you will be given cyclophosphamide by a continuous injection (using the catheter) for 2 days. You may also receive antibiotics, fluids, and other medications if your doctor feels it is necessary.

After you receive the chemotherapy, you will be given your treated bone marrow or blood stem cells back. To help speed up the recovery of white blood cells, you will also be given G-CSF by injection under the skin once a day until the white blood count has recovered (usually 2 to 3 weeks) and GM-CSF under the skin for a month. You may also receive antibiotics, fluids, and other medications if your doctor feels it is necessary. Blood tests (about 4 teaspoons) are repeated several times per week until blood counts are fully recovered and any side effects of the high dose therapy have resolved.

You will have check-up visits 1, 3, 6, and 12 months after the transplant. At these visits, you will have bone marrow samples collected to monitor the disease response. Bone marrow samples may also be collected for research at the same time points. These samples will be used to determine the survival of stem cells in laboratory conditions after the transplant. You will have blood collected (1- 4 tablespoons) for routine blood tests.

This is an investigational study. Busulfan, cyclophosphamide, G-CSF and GM-CSF are commercially available drugs. Up to 48 patients will take part in this study. All will be treated at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Philadelphia (Ph) chromosome positive CML < age 65 and older than 21 years.
* Ph positive CML that is either in: 1. late 1st chronic phase (> 2 years from diagnosis) 2. early chronic phase who did not achieve complete cytogenetic remission after one year on imatinib 3. beyond first chronic phase 4. accelerated phase 5. blastic phase that has responded to therapy (characterized by the presence of < 10% bone marrow and/or circulating blasts at consent signing) 6. chronic phase, developing imatinib resistance (loss of molecular remission defined as at least a 1 log increase in the BCR-ABL/ABL ratio, in 2 time points at least 1 month apart, or loss of cytogenetic remission)
* Patients must have a Zubrod PS < 3. Creatinine < 1.8 mg/dl
* Serum bilirubin </= 1.5 mg/dl
* Serum glutamate pyruvate transaminase (SGPT) < 3 x normal values
* Patients with an HLA identical sibling are eligible if they refuse allogeneic transplantation, or if they are ineligible for allogeneic transplantation due to age.
* DLCO >/= 50% of predicted
* Cardiac Ejection fraction >/= 40%

Exclusion Criteria:

* Uncontrolled life-threatening infections or comorbid condition that could impair tolerance to the regimen.
* HIV positivity.
* Pregnant or lactating women.
* CML in blastic phase that has not responded to therapy given prior to enrollment in this study (characterized by the presence of more than 9% bone marrow and/or peripheral blood blasts at the time of consent signing)
* Hepatitis B or C virus infection. Hepatitis B infection defined by positive DNA test, positive E and / or surface antigen.
* CML in first molecular remission.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-03; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Time to absolute neutrophil count (ANC) recovery to 500 | 30 Days
Survival Time | 30 Days (Success Rate + ANC Recovery to 500)

CONTACTS AND LOCATIONS:
Overall Officials: Marcos de Lima, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org